CLINICAL TRIAL: NCT06190444
Title: A Study of E-health Literacy in Athletes
Brief Title: E-health Literacy in Athletes
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Other Study IDs: KaratayUH11
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
e-health literacy in athletes is very important. The aim of this study was to determine the level of e-health literacy in athletes and to examine the relationship between age, gender, sports branches and injury sites.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the training,
* being an athlete for at least 2 years.

Exclusion Criteria:

* having any vision and hearing problems

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Athletes
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
E-health literacy | Baseline
  The E-Health Literacy Scale will used to determine the participants' e-health literacy.The scale consists of 2 items related to internet use and 8 items measuring internet attitude. The scale items are organized as "1= strongly disagree, 2= disagree, 3= undecided, 4= agree, 5= strongly agree" with a 5-point Likert-type scaling method. The lowest score is 8 points and the highest score is 40 points. A high score obtained from the scale indicates a high level of e-health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided